CLINICAL TRIAL: NCT04057781
Title: Pain and Neck Dysfunction Following Dry Needling With and Without Intramuscular Electrical Stimulus With 6 Week Follow Up
Brief Title: Pain and Neck Dysfunction Following Dry Needling With and Without Intramuscular Electrical Stimulus.
Acronym: DNvDNES-2019
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mary Hardin-Baylor (Other)
Responsible Party: Principal Investigator, Kindyle Brennan, Associate Professor, Doctor of Physical Therapy Program, University of Mary Hardin-Baylor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNvDNES-2019
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Neck Pain; Shoulder Pain; Myofascial Pain
MeSH Terms: conditions — Neck Pain; Shoulder Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Experimental There will be three groups in this study; control, DN alone and DN/IES. Each group will have approximately 20 subjects, resulting in approximately 60 subjects total. Subjects will be randomized into one of the three groups via block randomization method based on order of entry into the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention)
- Dry Needling (DN) (Active Comparator): Subjects will receive dry needling treatment every 2 weeks for 6 weeks (weeks 0, 2, 4, 6).
  Outcomes will be measured at baseline (week 0), 4 weeks after initiation of study (week 4), 6 weeks after initiation of study (week 6), and 6 weeks after last treatment (week 12).
  Interventions: Procedure: Dry Needling (DN)
- Dry Needling with Intramuscular ES (DNES) (Active Comparator): Subjects will receive dry needling treatment with electrical stimulation every 2 weeks for 6 weeks (week 0, 2, 4, 6)
  Outcomes will be measured at baseline (week 0), 4 weeks after initiation of study (week 4), 6 weeks after initiation of study (week 6), and 6 weeks after last treatment (week 12).
  Interventions: Procedure: Dry needling with Intramuscular electrical stimulation (DNES)

INTERVENTIONS:
Procedure: Dry Needling (DN) — One to three filament needles (similar to an acupuncture needle) with no medication will be inserted into the trigger point(s) of the muscle. The needles will be repositioned a few times to make the muscle twitch (local twitch response). After several twitches occur, the researcher will leave the needles as they are, and the subject will lie on a treatment table without moving arms or head, for 10 minutes. After 10 minutes the needles are removed and discarded.
  Arms: Dry Needling (DN)
Procedure: Dry needling with Intramuscular electrical stimulation (DNES) — One to three filament needles (similar to an acupuncture needle) with no medication will be inserted into the trigger point(s) of the muscle. The needles will be repositioned a few times to make the muscle twitch (local twitch response). After several twitches occur, the researcher will leave the needles as they are, and attach alligator clips to the needles to provide electrical stimulus for 10 minutes while the subject lies on a treatment table without moving arms or head. After 10 minutes, the electrical stimulus will be turned off and detached, and the needles removed and discarded.
  Arms: Dry Needling with Intramuscular ES (DNES)

SUMMARY:
Participants will be 18-59 years old who are recruited through a convenience sample from the UMHB/Belton community. There will be a randomized control trial consisting of three groups. Each participant will be assigned based on their order of entry to the study group assignment and then randomly organized via computer generation into 3 groups of 20 participants including a control group, a dry needling group (DN), and a dry needling E-stim group (DN-ES), resulting in approximately 60 total participants. Participants in the DN and DN-ES groups will be treated four times; at weeks 0, 2, 4 and 6 of the study. Data will be collected at weeks 4, 6 and 12 in all groups.

DETAILED DESCRIPTION:
Interventions per group:

Control: none

DN: 20-30 seconds of DN per trigger point in each involved trapezius muscle, needles rest in situ 10 min, needles removed.

DN-ES: 20-30 seconds of DN per trigger point (TrP) in each involved trapezius muscle, DC ES attached to needles crossing the most reactive TrP and current set to strong, but comfortable intensity at 10 MHz for 10 min, needles removed.

ELIGIBILITY:
Inclusion Criteria:

1. 18-59 years old
2. have an active email account
3. have at least one palpable active trigger point (TrP) (located in one or both upper trapezius)
4. English speaking

Exclusion Criteria:

1. current treatment or diagnosis related to cancer
2. active local or systemic infection
3. neurologic deficit
4. cognitive deficit
5. pregnancy
6. connective tissue disease and/or autoimmune disorder
7. tobacco use
8. received previous DN treatments within 6 weeks of the study,
9. experienced unilateral or bilateral neck/shoulder pain continuously for 3 months or longer
10. Neck Disability Index score < 6
11. Numerical Pain Rating Scale score < 3

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Change in numerical pain rating scale (NPRS)between groups | 6 weeks
  Between group difference in within group pain changes. The NPRS is an 11 point (0-10) scale with 10 meaning "the worst imaginable pain" and 0 meaning "no pain". It is reported as a whole number out of 10, and multiple ratings, i.e. worst, average, and best pain scores over the past 48 hours, can be averaged and reported as a single score.
Change in Neck Disability Index (NDI) | 6 weeks
  Between group difference in within group disability changes. The NDI is a questionnaire with 10 items including personal care, pain, reading, lifting, headaches, concentration, sleeping, work, driving, and recreation. Each section is scored on a 0 to 5 rating scale. Zero means 'No pain' and 5 means 'Worst imaginable pain'. Al the points can be summed to a total score. The test can be reported as a raw score, with a maximum score of 50, or as a percentage.

SECONDARY OUTCOMES:
Maintenance of improvement in pain scores (NPRS) | Compare 6 week data to 12 week data
  Difference between pain scores in both groups between the 6th week of weekly treatment and those 6 weeks after cessation of treatment. Scale is 11 points (0-10) with 10 being "the Analysis of within group pain scores. The NPRS is an 11 point (0-10) scale with 10 meaning "the worst imaginable pain" and 0 meaning "no pain". It is reported as a whole number out of 10, and multiple ratings, i.e. worst, average, and best pain scores over the past 48 hours, can be averaged and reported as a single score.
Maintenance of improvement in disability (NDI) | Compare 6 week data to 12 week data
  Difference between neck disability scores in both groups between the 6th week of weekly treatment and those 6 weeks after cessation of treatment. Between group difference in Analysis of within group disability changes. The NDI is a questionnaire with 10 items including personal care, pain, reading, lifting, headaches, concentration, sleeping, work, driving, and recreation. Each section is scored on a 0 to 5 rating scale. Zero means 'No pain' and 5 means 'Worst imaginable pain'. Al the points can be summed to a total score.
  Difference between neck disability scores in both groups between the 6th week of weekly treatment and those 6 weeks after cessation of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mary Hardin-Baylor, Belton, Texas, United States

IPD SHARING:
Plan to Share IPD: No